CLINICAL TRIAL: NCT05352711
Title: Effect of Virtual Reality Exercise on Pain and Range of Motion in Pediatrics With Second Degree Anterior Shoulder Burn Injuries
Brief Title: Virtual Reality on Pain and Range of Motion on Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Alaa Eid Abd-Elhafez, lecturer assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003467
Record Dates: First submitted 2022-04-13; First posted 2022-04-29 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Burns
Keywords: burn injuries
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active assisted exercise with Oculus Quest virtual reality (VR) group (Experimental): This group includes 30 patients suffered from pain and loss of shoulder flexion ROM, The patients will treated with active assisted exercise and with fully immersive Head-Mounted Display virtual reality ( Oculus Quest virtual reality (VR) headset with hand controller ) for 30 min. 2 times per week for 4 weeks The ROM will be assessed by mobile goniometer application and Smart phone version of visual analogue scale (VAS) to assess pain and The Quality-of-Life Scale for Children to assess the psychometric properties after the 1st session, day 14 and day 28.
  Interventions: Device: active assisted exercise and with fully immersive Head-Mounted Display virtual reality ( Oculus Quest virtual reality (VR) headset with hand con
- active assisted range of motion exercise group (Active Comparator): This group includes 30 patients suffering from pain and loss of shoulder flexion ROM. Patients will recieve active-assisted ROM physical therapy 2 sessions per week for 4 weeks.
  Interventions: Other: active assisted range of motion exercise

INTERVENTIONS:
Device: active assisted exercise and with fully immersive Head-Mounted Display virtual reality ( Oculus Quest virtual reality (VR) headset with hand con — VR is mainly created by generating visual effects through head-mounted display (HMD) systems. An HMD is a device worn on the head or as part of a helmet with a built-in display and lenses, allowing the user to experience the virtual world with the help of a wide viewing angle, head and hand movements tracking as well as objects interacting by controllers.
  Arms: active assisted exercise with Oculus Quest virtual reality (VR) group
Other: active assisted range of motion exercise — Patients were treated active assisted ROM physical therapy 2 sessions per week for 4 weeks.
  Arms: active assisted range of motion exercise group

SUMMARY:
The Purpose of the study is to determine the effect of virtual reality exercise on pain and shoulder range of motion in pediatrics with 2nd-degree anterior shoulder burn injuries.

DETAILED DESCRIPTION:
Burns are an important cause of injury to young children, being the third most frequent cause of injury resulting in death behind motor vehicle accidents and drowning. Burn injuries account for the greatest length of stay of all hospital admissions for injuries and costs associated with care are substantial. The majority of burn injuries in children are scald injuries resulting from hot liquids, occurring most commonly in children aged 0-4 years. Other types of burns include electrical, chemical and intentional injury. Mechanisms of injury are often unique to children and involve exploratory behavior without the requisite comprehension of the dangers in their environment.

Immersive virtual reality (VR) is a new form of cognitive distraction and has been found to be an effective adjunctive, nonpharmacologic analgesic for postburn physical therapy. The VR gives the individual the illusion of "going into" the 3-dimensional computer generated environment, as if it were a place in which they are actually physically present. The strength of the presence is thought to reflect the amount of attention that is drawn into the virtual world. Because VR is a highly attention-grabbing experience, it can be an effective psychological pain control technique. Less attention to pain can result in reductions in pain intensity, unpleasantness, and the amount of time patients spend thinking about their pain.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 9-16 years.
* Both sexes will participate in the study.
* Patients who suffered from anterior shoulder burns with involvement of axillary fold.
* patient who suffered from second degree burns.
* all patients are acute cases .

Exclusion Criteria:

* injuries to the face or head
* Injuries in hands
* Cognitive impairment
* A history of severe motion sickness
* Mental health problems.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
status of ROM for shoulder flexion assessment in day 1 | Goniometer record apps was used to measure shoulder flexion range of movement (ROM) in day 1
  mobile applications (apps) specifically designed to measure ROM
change of ROM for shoulder flexion assessment in day 14 | Goniometer record apps was used to measure shoulder flexion range of movement (ROM) in day 14
  mobile applications (apps) specifically designed to measure ROM
change of ROM for shoulder flexion assessment in day 28 | Goniometer record apps was used to measure shoulder flexion range of movement (ROM) in day 28
  mobile applications (apps) specifically designed to measure ROM
status of shoulder pain assessment in day 1 | evaluate psychometric properties within the distinct targeted samples in day 1
  Smart phone version of visual analogue scale (VAS) for assessing the pain ,the user touches the line, marking the location along the line that indicates the severity of the pain. An integer score between 0 and 100 is calculated based on the location of the marker relative to the ends of the line.(0 indicates no pain while 100 indicates worest pain)
change of shoulder pain assessment in day 14 | evaluate psychometric properties within the distinct targeted samples in day 14
  Smart phone version of visual analogue scale (VAS) for assessing the pain ,the user touches the line, marking the location along the line that indicates the severity of the pain. An integer score between 0 and 100 is calculated based on the location of the marker relative to the ends of the line.(0 indicates no pain while 100 indicates worest pain)
change of shoulder pain assessment in day 28 | evaluate psychometric properties within the distinct targeted samples in day 28
  Smart phone version of visual analogue scale (VAS) for assessing the pain ,the user touches the line, marking the location along the line that indicates the severity of the pain. An integer score between 0 and 100 is calculated based on the location of the marker relative to the ends of the line. (0 indicates no pain while 100 indicates worest pain)

SECONDARY OUTCOMES:
presentation of an individual's perception of their current health state | questionnaire is used to asses the quality of patient's life at the first day of treatment
  Quality-of-Life Scale from 0 to 10 (0 is the worst health you could imagine. 10 is the best health you could imagine)
change in presentation of an individual's perception of their current health state | this questionnaire will be used to asses the quality of patient's life at the day 28 of treatment
  Quality-of-Life Scale from 0 to 10 (0 is the worst health you could imagine. 10 is the best health you could imagine)

CONTACTS AND LOCATIONS:
Overall Officials: Amal Mohamed Abd Albaky, Professor, Study Chair — Vice dean of high education Faculty of Physical Therapy Cairo University
Locations (1):
- Ahmed Orabi hospital for burn and tumors, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided